CLINICAL TRIAL: NCT05405985
Title: A Randomized, Single-Dose, Open-Label, Parallel-Group Study in Healthy Volunteers to Assess the Relative Bioavailability of a Subcutaneous Dose of Nemolizumab When Administered With Auto-Injector Compared to Dual-Chamber Syringe
Brief Title: Study to Access the Relative Bioavailability of Subcutaneous Dose of Nemolizumab When Administered Via Auto-Injector Versus Dual-Chamber Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.201590
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Auto-Injector (AI); Dual-Chamber Syringe (DCS); Atopic dermatitis (AD); Prurigo nodularis (PN)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab With Auto-Injector (AI) (Experimental): Participants received a 60 milligrams (mg) dose of nemolizumab as 2 successive subcutaneous (SC) injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 centimeters [cm]) apart with AI on Day 0 (injection day).
  Interventions: Drug: Nemolizumab
- Nemolizumab With Dual Chamber Syringe (DCS) (Experimental): Participants received a 60-mg dose of nemolizumab as 2 successive subcutaneous injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with DCS on Day 0 (injection day).
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Nemolizumab — Nemolizumab with Auto-Injector (AI).
  Arms: Nemolizumab With Auto-Injector (AI)
Drug: Nemolizumab — Nemolizumab with Dual-Chamber Syringe (DCS).
  Arms: Nemolizumab With Dual Chamber Syringe (DCS)

SUMMARY:
This study was to compare the rate and extent of absorption of a single dose of nemolizumab administered with auto-injectors [AI] (test) versus dual-chamber syringes [DCS] (reference) under controlled conditions in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 65 years at screening visit.
* Body weight >= 45 kilogram (kg) and body mass index between >=18.0 and <30.0 kilograms per meter squared (kg/m^2) at both screening and baseline visits.
* Medically healthy with normal clinical status as judged by the investigator based on medical history, physical examination, and clinical laboratory tests.
* Willing to abstain from all prescription medications during the study, (defined hereafter as after signing of informed consent form), except to treat AEs and contraception, and as permitted under Exclusion 2. Limited use of non-prescription medications/supplements that were not believed to affect participant's safety or the overall results of the study might be permitted at the discretion of investigator.
* Female participants of childbearing potential (i.e., fertile, after menarche and, until becoming postmenopausal unless permanently sterile) must agree either to be strictly abstinent throughout the study and for 12 weeks after the study drug injection, or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the study drug injection. Males are not required to use contraception, and there is no restriction on sperm donation.
* Female participants of non-childbearing potential must meet one of these criteria; absence of menstrual bleeding for 1 year before the screening visit with no other medical reason, confirmed with follicle-stimulating hormone (FSH) level in the postmenopausal range or documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before the study.
* Willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol.
* Understood and signed an informed consent form before any investigational procedure(s) are performed.

Exclusion Criteria:

* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, e.g., monoclonal antibody) or to any of the study drug excipients.
* Cutaneous infection within 1 week before the baseline visit or any infection requiring treatment with oral, parental antibodies, antivirals, antiparasitics, or antifungals within 2 weeks before the baseline visit.
* Any confirmed or suspected coronavirus disease (COVID-19) infection within 2 weeks before screening or baseline visit.
* Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], hepatitis C [HCV] antibody with positive HCV RNA, or human immunodeficiency virus [HIV] antibody) at the screening visit.
* Known or suspected immunosuppression or unusually frequent, recurrent, severe, or prolonged infections as per investigator judgment.
* History of lymphoproliferative disease or history of malignancy of any organ system within last 5 years, except for basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that have been treated and have no clinical evidence of recurrence in the last 12 weeks before baseline visit, or actinic keratoses that have been treated.
* Previous treatment with Nemolizumab.
* Known active or untreated latent tuberculosis infection.
* Any condition that may interfere with study assessments (e.g., poor venous access or needle phobia).
* Having received a live-attenuated or non-live vaccine within 4 weeks before the baseline visit or are expected to be vaccinated during the study or during the 12 weeks after the last study drug injection, except for non-live seasonal vaccinations, COVID-19 and /or emergency vaccinations.
* Planned or expected major surgical procedure during the clinical study.
* Pregnant women, breastfeeding women, or women planning a pregnancy during the study or 12 weeks after the study drug injection.
* Participating or participated in any other study with an investigational drug or device within the past 8 weeks before the screening visit, or is in an exclusion period from a previous study.
* Participants who have donated ≥ 500 mL of blood in the last 3 months before doing.
* History of alcohol or substance abuse within 6 months of the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Galderma Investigational Site 7024, Tempe, Arizona
  - Galderma Investigational Site 7023, Lincoln, Nebraska

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites in United States from 11 August 2022 to 08 December 2022.
Pre-assignment Details: A total of 192 participants were randomized in two treatment group. 96 participants received nemolizumab with auto-injector (AI) and remaining 96 participants received nemolizumab with dual chamber syringe (DCS).
Groups:
- Nemolizumab With Dual Chamber Syringe (DCS): Participants received a 60-mg dose of nemolizumab as 2 successive SC injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with DCS on Day 0 (injection day).
Period: Overall Study
Arm/Group | Nemolizumab With Auto-Injector (AI) | Nemolizumab With Dual Chamber Syringe (DCS)
Started | 96 | 96
Completed | 95 | 96
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all randomized participants who received the single dose of nemolizumab and was the primary population for all safety data.
Groups:
- Nemolizumab With AI: Participants received a 60 mg dose of nemolizumab as 2 successive SC injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with AI on Day 0 (injection day).
- Nemolizumab With DCS: Participants received a 60-mg dose of nemolizumab as 2 successive SC injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with DCS on Day 0 (injection day).
- Total: Total of all reporting groups
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS | Total
Number analyzed (Participants) | 96 | 96 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.71) | 42.1 (12.52) | 41.5 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 62 | 117
  Male | 41 | 34 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 51 | 104
  Not Hispanic or Latino | 43 | 45 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 82 | 80 | 162
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Nemolizumab
Description: Cmax was defined as the observed maximum serum concentration of nemolizumab. Cmax was used to measure the rate of absorption of nemolizumab.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22, 29, 36, 43, 50, 57, 71, and 85 post-dose
Population: Analysis was performed on pharmacokinetics (PK) population which included all randomized participants who received the dose of nemolizumab and provided evaluable data that can be used for the PK analyses.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 96 | 96
micrograms per milliliter (mcg/mL) | 8.00 (2.34) | 7.51 (2.31)

2. Primary Outcome: Area Under Concentration-time Curve Extrapolated to Infinity (AUC0-inf) of Nemolizumab
Description: AUC0-inf was defined as area under the plasma concentration-time curve from time 0 to infinity according to the equation: AUC0-inf = AUClast + Clast/λz; where λz = slope of the regression line of the terminal phase of the plasma concentration versus time curve, in semi-logarithmic scale; and Clast = last measurable drug concentration.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22, 29, 36, 43, 50, 57, 71, and 85 post-dose
Population: Analysis was performed on PK population which included all randomized participants who received the dose of nemolizumab and provided evaluable data that can be used for the PK analyses. Here, 'overall number of participants analyzed, N' signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms*day per milliliter
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 95 | 96
micrograms*day per milliliter | 270 (85.8) | 279 (89.7)

3. Secondary Outcome: Area Under the Concentration-time Curve Over the Specified Interval (AUC0-4 Weeks) of Nemolizumab
Description: AUC0-4 weeks was defined as area under the concentration-time curve from time 0 to 4 weeks after study drug administration calculated with the linear trapezoidal method.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22 and 29 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrograms*day per milliliter
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 95 | 96
micrograms*day per milliliter | 157 (37.9) | 155 (39.8)

4. Secondary Outcome: Area Under Concentration-time Curve From Administration to the Last Observed Concentration Time t (AUC0-last) of Nemolizumab
Description: AUC0-last was defined as area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22, 29, 36, 43, 50, 57, 71, and 85 post-dose
Population: Analysis was performed on PK population which included all randomized participants who received the dose of nemolizumab and provided evaluable data that can be used for the PK analyses.
Measure: Mean (Standard Deviation); unit: micrograms*day per milliliter
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 96 | 96
micrograms*day per milliliter | 250 (73.6) | 260 (75.4)

5. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Nemolizumab
Description: Tmax was defined as the time taken to reach the maximum observed serum concentration.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22, 29, 36, 43, 50, 57, 71, and 85 post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 96 | 96
days | 4.99 [1.00 to 21.99] | 5.99 [1.00 to 22.00]

6. Secondary Outcome: Half-life (t1/2) of Nemolizumab
Description: t1/2 is defined as time required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose, 12 hours, 24 hours, Days 3, 4, 5, 6, 7, 8, 9, 10, 11, 15, 22, 29, 36, 43, 50, 57, 71, and 85 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 95 | 96
days | 18.0 (5.91) | 18.5 (4.52)

7. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) Response Against Nemolizumab
Description: ADA positive was defined as a sample that was evaluated as positive in both the ADA screening and confirmatory assays. ADA positive participants was defined as participants who had at least 1 positive ADA result.
Time Frame: Pre-dose, Day 29 and 85 post-dose
Population: Analysis was performed on safety population that included all randomized participants who received the single dose of nemolizumab and was the primary population for all safety data. Here, 'overall number of participants analyzed, N' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
Number analyzed (Participants) | 95 | 96
Participants
  Pre-dose: ADA postive | 6 | 8
  Day 29: ADA positive | 2 | 4
  Day 85: ADA positive | 2 | 8

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 12
Description: Analysis was performed on safety population that included all randomized participants who received the single dose of nemolizumab and was the primary population for all safety data.
Groups:
- Nemolizumab With AI: Participants received a 60 mg dose of nemolizumab as 2 successive SC injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with AI on Day 0.
- Nemolizumab With DCS: Participants received a 60-mg dose of nemolizumab as 2 successive SC injections of 30 mg nemolizumab at either of the same location i.e., abdomen, front upper thigh, or outer upper arm and on the same side with injection sites at least 1 inch (2.5 cm) apart with DCS on Day 0.
Arm/Group | Nemolizumab With AI | Nemolizumab With DCS
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 41/96 | 54/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab With AI (N=96) | Nemolizumab With DCS (N=96)
Palpitations (Cardiac disorders) | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip pruritus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Palatal disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Hunger (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 2
Injection site erythema (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 0
Injection site pruritus (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Procedural failure (General disorders) | 1 | 0
Vaccination site pain (General disorders) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Heart rate increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 1
Weight increased (Investigations) | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 8 | 22
Migraine (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Procedural anxiety (Psychiatric disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 2
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT05405985/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05405985/SAP_001.pdf